CLINICAL TRIAL: NCT03124290
Title: The Effect of Attention Distractor During Cardiopulmonary Resuscitation on the Quality of Chest Compression: Randomized Crossover Trial With Simulated Situation
Brief Title: The Effect of Attention Distractor on the Quality of Chest Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Joon Min Park, Assistant Professor, Inje University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2017-04-007
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Cardiopulmonary Resuscitation, Simulation Training
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPR with attention distraction first (Other): First, they perform two-minute chest compressions with conducting the PASAT. After 20 mins' rest, they perform two-minute chest compressions without conducting the PASAT.
  Interventions: Other: paced auditory serial addition test (PASAT)
- CPR without attention distraction first (Other): First, they perform two-minute chest compressions without conducting the PASAT. After 20 mins' rest, they perform two-minute chest compressions with conducting the PASAT.
  Interventions: Other: paced auditory serial addition test (PASAT)

INTERVENTIONS:
Other: paced auditory serial addition test (PASAT) — A number between 1 to 9 is called every three seconds through a speaker, and the performer calculates the last two numbers and shouts the answer.

SUMMARY:
The investigators plan to investigate the effect of attention distractor on the quality of chest compression during cardiopulmonary resuscitation. For this, a simulated study with Manikin is performed and the paced auditory serial addition test (PASAT) is used for distracting performer's attention.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers who completed basic life support course among medical personnel (doctors, nurses, paramedics) working in a university hospital

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-05-14 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
adequate compression rate | two minutes
  the percentage of chest compression with adequate rate (100-120 per minute) during two-minute chest compression. Formula(%)=number of adequate chest compressions (rate:100-120/min) x 100 / number of all chest compressions during two minutes

SECONDARY OUTCOMES:
adequate compression depth | two minutes
  the percentage of chest compression with adequate depth (5-6cm) during two-minute chest compression. Formula(%)= number of adequate chest compressions(depth=5-6cm)x 100 / all chest compressions during two minutes
adequate chest recoil | two minutes
  the percentage of chest compression with adequate chest recoil during two-minute chest compression. Formula(%)=number of adequate chest recoils(automatically measured with simulator) x 100/ number of all chest compressions during two minutes
mean compression rate | two minutes
  Average of compression rate during two-minute chest compression. The scale for this outome is 'number per minute'.
mean compression depth | two minutes
  Average of compression depth during two-minute chest compression. The scale for this outcome is 'cm'.
Subjective difficulty | Two minutes
  Each performer rate the subjective difficulties of two arms with the 100mm VAS (0: very easy, 100: very difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Min Park, Principal Investigator — Inje University Ilsan Paik Hospital
Locations (1):
- Inje University Ilsan Paik Hospital, Goyang-si, South Korea

REFERENCES:
- [Derived] Lee K, Kim MJ, Park J, Park JM, Kim KH, Shin DW, Kim H, Jeon W, Kim H. The effect of distraction by dual work on a CPR practitioner's efficiency in chest compression: A randomized controlled simulation study. Medicine (Baltimore). 2017 Oct;96(43):e8268. doi: 10.1097/MD.0000000000008268. PMID 29068995